CLINICAL TRIAL: NCT04392141
Title: Application of Colchicine Plus Herbal Phenolic Monoterpene Fractions to Treat COVID-19
Brief Title: Colchicine Plus Phenolic Monoterpenes to Treat COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kermanshah University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Ali Mostafaie, PhD, Professor of Immunology, Kermanshah University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1399.062
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19; Colchicine; Phenolic Monoterpenes
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Experimental): Patients diagnosed with COVID-19 which receive the standard treatment national guideline
  Interventions: Drug: Standard Treatment
- Colchicine and Herbal Phenolic Monoterpene Fractions (Experimental): Patients diagnosed with COVID-19 which receive the standard treatment national guideline plus Colchicine and Herbal Phenolic Monoterpene Fractions
  Interventions: Drug: Oral administration of Colchicine plus Herbal Phenolic Monoterpene Fractions

INTERVENTIONS:
Drug: Standard Treatment — Standard Treatment for COVID-19 based on National Recommendations
  Arms: Standard Treatment
Drug: Oral administration of Colchicine plus Herbal Phenolic Monoterpene Fractions — Colchicine plus a Herbal extraction containing a Phenolic Monoterpene Fractions will be added to standard treatment in patients with COVID-19.
  Arms: Colchicine and Herbal Phenolic Monoterpene Fractions

SUMMARY:
In this randomized controlled clinical trial, defined cases of COVID-19 with mild, moderate, or severe pneumonia (according to the NIH guideline) were treated with conventional treatment regimens (controls) as well as in combination with oral administration of colchicine plus herbal phenolic monoterpene fractions (intervention arm). After randomization, each group received the mentioned treatments and were evaluated for different variables including mortality, hospitalization duration, intensive care unit (ICU) administration ratios as well as laboratory variables such as leukocytes and lymphocytes count. The follow-up period considered as 2 weeks after discharge. The mentioned variables were assessed as before and after receiving the treatment in each group as well as intergroup analysis for comparing both baseline and final values.

ELIGIBILITY:
Inclusion Criteria:

* Defined cases of COVID-19 based on laboratory and/or radiological and clinical manifestation

Exclusion Criteria:

* Age <10, Pregnancy, Sever kidney dysfunction, Previous history of allergy to Colchicine, not willing to sign informed consent form

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mostafaie, PhD, Principal Investigator — Medical Biology Research Center, Kermanshah University of Medical Sciences, Kermanshah, Iran.
Locations (1):
- Medical Biology Research Center, Kermanshah University of Medical Sciences, Kermanshah, Iran, Kermanshah, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nerlekar N, Beale A, Harper RW. Colchicine--a short history of an ancient drug. Med J Aust. 2014 Dec 11;201(11):687-8. doi: 10.5694/mja14.00846. No abstract available. PMID 25495322
- [Background] Larsson S, Ronsted N. Reviewing Colchicaceae alkaloids - perspectives of evolution on medicinal chemistry. Curr Top Med Chem. 2014;14(2):274-89. doi: 10.2174/1568026613666131216110417. PMID 24359194
- [Background] Slobodnick A, Shah B, Krasnokutsky S, Pillinger MH. Update on colchicine, 2017. Rheumatology (Oxford). 2018 Jan 1;57(suppl_1):i4-i11. doi: 10.1093/rheumatology/kex453. PMID 29272515
- [Background] Cronstein BN, Molad Y, Reibman J, Balakhane E, Levin RI, Weissmann G. Colchicine alters the quantitative and qualitative display of selectins on endothelial cells and neutrophils. J Clin Invest. 1995 Aug;96(2):994-1002. doi: 10.1172/JCI118147. PMID 7543498
- [Background] Umar S, Shah MAA, Munir MT, Yaqoob M, Fiaz M, Anjum S, Kaboudi K, Bouzouaia M, Younus M, Nisa Q, Iqbal M, Umar W. RETRACTED: Synergistic effects of thymoquinone and curcumin on immune response and anti-viral activity against avian influenza virus (H9N2) in turkeys. Poult Sci. 2016 Jul 1;95(7):1513-1520. doi: 10.3382/ps/pew069. Epub 2016 Mar 4. PMID 26944958
- [Background] Wu QF, Wang W, Dai XY, Wang ZY, Shen ZH, Ying HZ, Yu CH. Chemical compositions and anti-influenza activities of essential oils from Mosla dianthera. J Ethnopharmacol. 2012 Jan 31;139(2):668-71. doi: 10.1016/j.jep.2011.11.056. Epub 2011 Dec 16. PMID 22193174
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: Year] | 54.11 (14.39) | 52.99 (15.88) | 53.55 (15.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 33 | 32 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iran | 60 | 60 | 120
Hypertension [Count of Participants; unit: Participants] | 12 | 20 | 32
Diabetic mellitus [Count of Participants; unit: Participants] | 3 | 6 | 9
Malignancy [Count of Participants; unit: Participants] | 2 | 5 | 7
Autoimmune diseases [Count of Participants; unit: Participants] | 3 | 6 | 9
Smoking/Substance abuse [Count of Participants; unit: Participants] | 2 | 8 | 10
Severe to critically ill COVID-19 [Count of Participants; unit: Participants] — Moderate Illness: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have saturation of oxygen (SpO2) ≥94%.
  Severe Illness: Individuals who have SpO2 <94%, respiratory frequency >30 breaths/min, or lung infiltrates >50%.
  Critical Illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction.
  The definition of severe to critically ill COVID-19 patient is according to the National Health Institute (NIH).
  Participants | 48 | 52 | 100
lymphocytes count [Mean (Standard Deviation); unit: cells*1000/mm^3] | 1.19 (0.45) | 1.31 (0.64) | 1.26 (0.56)
LDH [Mean (Standard Deviation); unit: U/L] | 664.98 (295.84) | 680.27 (471.44) | 674.20 (401.78)
SpO2 [Mean (Standard Deviation); unit: Percentage of O2 saturation] | 87.39 (6.32) | 90.94 (3.27) | 89.53 (4.48)

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rate
Description: All cause of death in duration hospitalization
Time Frame: From admission to 14 days after being discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
Number analyzed (Participants) | 60 | 60
Participants | 6 | 1
Statistical Analysis 1: Comparison: Standard Treatment vs Colchicine and Herbal Phenolic Monoterpene Fractions; Test type: Equivalence — equivalence of odds of death between both groups; p = 0.0318, Fisher Exact; Odds Ratio (OR) = 9.87, 95% CI 2-sided [1.16 to 83.89]

2. Secondary Outcome: SpO2
Description: Change in patients' oxygen saturation levels assessed by non-invasive method (pulse oximetry)
Time Frame: Admission to discharge dates (approximately 4-14 days after admission). Discharge variables considered as the last available data before their death for the expired patients.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
Number analyzed (Participants) | 60 | 60
Percentage of oxygen saturation
  Admission | 87.39 (6.32) | 90.94 (3.27)
  Discharge | 92.89 (1.76) | 93.49 (2.12)
Statistical Analysis 1: Comparison: Standard Treatment; Statistical comparison of SpO2 (%) between admission and discharge times in standard treatment group; Test type: Equivalence — equivalence of SpO2 percentage between admission and discharge phases; p = 0.0001, t-test, 2 sided; Paired T-test; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-7.03 to -3.96]
Statistical Analysis 2: Comparison: Colchicine and Herbal Phenolic Monoterpene Fractions; Statistical comparison of SpO2 % between admission and discharge times in the Colchicine and Herbal Phenolic Monoterpene Fractions treatment; Test type: Equivalence — equivalence of SpO2 percentage between admission and discharge phases; p = 0.0001, t-test, 2 sided; Paired T-test; Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-3.28 to -1.81]

3. Secondary Outcome: Length of Hospitalization
Description: Day(s) each patient has spent in the hospital as an inpatient.
Time Frame: The duration of hospitalization for the patients (admission to discharge dates, approximately 4-14 days after admission). The patients who died were excluded.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
Number analyzed (Participants) | 54 | 59
Day | 6.39 (2.59) | 4.17 (1.34)
Statistical Analysis 1: Comparison: Standard Treatment vs Colchicine and Herbal Phenolic Monoterpene Fractions; Test type: Equivalence — equivalence of means of the length of hospitalization between both groups; p = 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.22, 95% CI 2-sided [1.63 to 2.80]

4. Secondary Outcome: Lymphocyte Count
Description: Lymphocyte count*1000/ mm^3
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells*1000/mm^3
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
Number analyzed (Participants) | 60 | 60
cells*1000/mm^3
  Admission | 1.19 (0.45) | 1.31 (0.64)
  Discharge | 1.17 (0.49) | 1.74 (0.83)
Statistical Analysis 1: Comparison: Standard Treatment; Statistical comparison of lymphocytes count between admission and discharge times in standard treatment; Test type: Equivalence — equivalence of mean of lymphocytes count between admission and discharge phases; p = 0.80, t-test, 2 sided; Paired T-test; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.136 to 0.176]
Statistical Analysis 2: Comparison: Colchicine and Herbal Phenolic Monoterpene Fractions; Statistical comparison of lymphocytes count between admission and discharge times in Colchicine and Herbal Phenolic Monoterpene Fractions treatment; Test type: Equivalence — equivalence of mean of lymphocytes count between admission and discharge phases; p = 0.0001, t-test, 2 sided; Paired T-test; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.63 to -0.23]

5. Secondary Outcome: Serum Lactate Dehydrogenase
Description: Serum lactate dehydrogenase: LDH (U/L)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
Number analyzed (Participants) | 60 | 60
U/L
  Admission | 664.98 (295.84) | 680.27 (471.44)
  Discharge | 691.04 (299.09) | 542.94 (225.67)
Statistical Analysis 1: Comparison: Standard Treatment; Statistical comparison of LDH between admission and discharge times in standard treatment; Test type: Equivalence — equivalence of mean of LDH between admission and discharge phases; p = 0.602, t-test, 2 sided; Paired T-test; Mean Difference (Final Values) = -26.06, 95% CI 2-sided [-124.76 to 72.64]
Statistical Analysis 2: Comparison: Colchicine and Herbal Phenolic Monoterpene Fractions; Statistical comparison of LDH between admission and discharge times in Colchicine and Herbal Phenolic Monoterpene Fractions treatment; Test type: Equivalence — equivalence of mean of LDH between admission and discharge phases; p = 0.006, t-test, 2 sided; Paired T-test; Mean Difference (Final Values) = 137.33, 95% CI 2-sided [38.19 to 236.46]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Standard Treatment | Colchicine and Herbal Phenolic Monoterpene Fractions
All-Cause Mortality (participants affected / at risk) | 6/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 2/60 | 4/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (N=60) | Colchicine and Herbal Phenolic Monoterpene Fractions (N=60)
Nausea with or without vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Restlessness (Nervous system disorders) | 0 (0) | 1 (1)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04392141/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04392141/SAP_001.pdf